CLINICAL TRIAL: NCT01988090
Title: A Randomized, Controlled Trial of High Dose vs. Standard Dose Vitamin D for Aromatase-Inhibitor Induced Arthralgia in Breast Cancer Survivors
Brief Title: High Dose Vitamin D vs Standard Dose Vitamin D Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: An interim analysis demonstrated no benefit of high dose vitamin D when compared to standard dose vitamin D in the reduction or prevention of arthralgia
Sponsor: Mothaffar Rimawi (Other)
Responsible Party: Sponsor-Investigator, Mothaffar Rimawi, Professor, Baylor Breast Care Center
Organization: Baylor Breast Care Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-33261
Record Dates: First submitted 2013-11-07; First posted 2013-11-20 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Hormone Receptor Positive; Vitamin D
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Dose Vitamin D ARM (Experimental): 50,000 IU Vitamin D supplement
  Interventions: Drug: 50,000 IU Vitamin D supplement
- 800 IU Vitamin D Supplement (Active Comparator): 800 IU Vitamin D Supplement
  Interventions: Drug: 800 IU Vitamin D Supplement

INTERVENTIONS:
Drug: 800 IU Vitamin D Supplement — Standard Dose
  Arms: 800 IU Vitamin D Supplement
Drug: 50,000 IU Vitamin D supplement — High Dose
  Arms: High Dose Vitamin D ARM

SUMMARY:
This study is being done to look at the difference, if there is a difference between two different doses of Vitamin D and the reduction of joint/muscle pain (arthralgia)that is caused by taking anti-estrogen medications (aromatase inhibitors) by breast cancer patients. The investigators hope to learn if taking a higher dose of Vitamin D is a good way to prevent aromatase inhibitor arthralgia (AIA).

DETAILED DESCRIPTION:
Treatments with anti-estrogen agents for hormone receptor positive breast cancer is the most efficacious of systemic therapies, with aromatase inhibitors (AI's) being considered the most active anti-estrogen therapy in early stage breast cancer. But, use of these treatments has been shown to cause musculoskeletal (joint/muscle) side effects that sometimes cause patients to discontinue the use of them. Also, Vitamin D deficiency is a well know cause of a wide array of musculoskeletal issues. There is evidence that Vitamin D supplementation may help prevent arthralgia while on AI's. Therefore, the investigators want to see if giving a higher dose of Vitamin D could decrease the incidence of AIA as compared to a standard dose of Vitamin D. The investigators believe that this could possibly result in patients continued treatment with AI therapy for hormone receptor positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be female and at least 21 years of age
* Signed informed consent
* Patients must have had histologically confirmed stage I-III breast carcinoma that is positive for Estrogen Receptor (ER) and/or Progesterone Receptor (PR).
* Post-menopausal
* Beginning adjuvant aromatase inhibitor therapy, with no previous use within the last 6 weeks
* Bisphosphonates are allowed at the treating investigator¡¦s discretion
* Performance status (WHO/ECOG scale) 0-2.

Exclusion Criteria:

* History of kidney stones
* Hypercalcemia at baseline, defined as any corrected calcium greater than the laboratory's normal parameters
* History of either symptomatic hypercalcemia or hyperparathyroidism, at the treating investigator's discretion
* Baseline Vitamin D level greater than 50 ng/mL
* Inability or unwillingness to comply with, or follow study procedures.
* Currently taking Phenytoin or phenobarbital -7 Currently taking cholestyramine or orlistat
* Malabsorption syndrome, such as Crohn's disease

Prohibited Therapies: Patients may not take additional Calcium and Vitamin D aside from the study medications. Patients who are on cholestyramine or orlistat will not be allowed on the trial. Also, patients who are taking phenytoin or phenobarbital are not allowed on the trial either because of interaction between Vitamin D and anti-epileptic medications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2018-07-21 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar Rimawi, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Washington University / Siteman Cancer Center, St Louis, Missouri
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Start Treament After Randomization
Arm/Group | High Dose Vitamin D ARM | 800 IU Vitamin D Supplement
Started | 46 | 47
Completed (Complete 12 weeks treatment) | 44 | 43
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Protocol Violation | 0 | 1
Period: Complete Study After Start
Arm/Group | High Dose Vitamin D ARM | 800 IU Vitamin D Supplement
Started | 44 | 43
Completed | 41 | 42
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Vitamin D ARM | 800 IU Vitamin D Supplement | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (7) | 63.8 (8.6) | 63.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 93
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 22 | 41
  Not Hispanic or Latino | 26 | 24 | 50
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 6 | 17
  White | 33 | 39 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 46 | 47 | 93
Serum 25-hydroxyvitamin D level [Mean (Standard Deviation); unit: ng/mL] | 21.7 (8.7) | 24.2 (7.1) | 23 (8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Aromatase Inhibitor Induced Arthralgia (AIA) After 12 Weeks of Therapy
Description: Aromatase Inhibitor Arthralgia (AIA) was assessed by a questionnaire that describe the level of pain experienced by the participant. The questionnaire asks 20 questions scored 0-3 in 8 categories of functioning: dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. An average composite score on the HAQ-II was calculated. The visual analog scale is the other major component of the HAQ-II, which we ask patients to mark where their pain lies on a horizontal line and we converts the number into a score from 0 to 3. For the purposes of this study, AIA will be defined as any of the following criteria: 1) increase in HAQ-II score from baseline by 0.2 or greater; or 2) increase in visual analog pain score by 0.3 or greater.
Time Frame: 12 weeks
Population: ITT population. All patients who were randomized in the study were included in the overall evaluation of response (intent-to-treat analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Vitamin D ARM | 800 IU Vitamin D Supplement
Number analyzed (Participants) | 46 | 47
Participants
  development of AIA | 25 | 27
  no development of AIA | 21 | 20
Statistical Analysis 1: Comparison: High Dose Vitamin D ARM vs 800 IU Vitamin D Supplement; Test type: Superiority; p = 0.7635, Chi-squared

2. Secondary Outcome: Compliance With Anti-Cancer Treatment
Description: We checked compliance of aromatase inhibitor therapy during the study by reviewing the patient's use of AI drug. This will be done by counting remaining pills in patient's bottles of AI at 52 weeks. A percentage of the number of pills were actually taken of the number of pills should be taken was calculated.
Time Frame: 52 Weeks
Population: Compliance was assessed at week 52. Only 14 patients have compete the data collection.
  Form was not completed due to not starting the treatment, or not finishing the treatment, or no source data.
Measure: Mean (Standard Deviation); unit: percentage of pills taken
Arm/Group | High Dose Vitamin D ARM | 800 IU Vitamin D Supplement
Number analyzed (Participants) | 6 | 8
percentage of pills taken | 0.981 (0.047) | 0.965 (0.07)

3. Secondary Outcome: Association Between Vitamin D Levels Changes and Treatment.
Description: Patients' serum 25-hydroxyvitamin D level were tested at baseline and week 12. The changes between baseline and week 12 were calculated.
Time Frame: 12 weeks
Population: Patients who had serum 25-hydroxyvitamin D level tested at baseline and week 12 were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | High Dose Vitamin D ARM | 800 IU Vitamin D Supplement
Number analyzed (Participants) | 39 | 36
ng/mL | 28.8 (14.5) | 5.2 (7.3)
Statistical Analysis 1: Comparison: High Dose Vitamin D ARM vs 800 IU Vitamin D Supplement; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

4. Other Pre Specified Outcome: Grip Strength
Description: Exploratory Endpoints For each patient on the study, grip strength will be correlated with AIA score using Spearman correlation at three time points throughout the study - baseline, week 12, and week 52.
Time Frame: 52 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 56 weeks. Adverse events experienced by participants were collected and reported from initiation of study medication, throughout the study (52 weeks treatment), and within 30 days of the last dose of study medication.
Arm/Group | High Dose Vitamin D ARM | 800 IU Vitamin D Supplement
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43
Serious Adverse Events (participants affected / at risk) | 2/44 | 0/43
Other Adverse Events (participants affected / at risk) | 35/44 | 36/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Vitamin D ARM (N=44) | 800 IU Vitamin D Supplement (N=43)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Vitamin D ARM (N=44) | 800 IU Vitamin D Supplement (N=43)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 6 (6) | 4 (4)
Pain (General disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (25) | 19 (22)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7)
headache (Nervous system disorders) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (12) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 4 (4) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
vaginal dryness (Reproductive system and breast disorders) | 5 (5) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hot flashes (Vascular disorders) | 23 (25) | 20 (22)
Hypertension (Vascular disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT01988090/Prot_SAP_000.pdf